CLINICAL TRIAL: NCT00126919
Title: Randomized Crossover Trial of Sonication Followed by 5 Minute LMX4 Application Compared With 30 Minute LMX4 Application for Topical Anesthesia Prior to Subcutaneous Port Access in Children
Brief Title: Reduction of Topical Anesthetic Time for Subcutaneous Port Access Using Ultrasound
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, William Zempsky, MD, Director, Pain Relief Program, Connecticut Children's Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05-002
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

INTERVENTIONS:
Device: SonoPrep

SUMMARY:
Children ages 3-17 who are undergoing port access receive both standard care, topical medicine for numbing (LMX4), and the study intervention which utilizes ultrasound to speed the onset of LMX4 from 30 minutes to 5 minutes. The procedures will be performed on 2 separate visits to the clinic. The child's pain with the access procedure is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3-17 with subcutaneous port

Exclusion Criteria:

* Emergent need for port access
* Allergy to lidocaine sodium lauryl sulfate

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2004-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
pain

SECONDARY OUTCOMES:
tolerability
safety-skin effects

CONTACTS AND LOCATIONS:
Overall Officials: William T. Zempsky, MD, Principal Investigator — CT Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States